CLINICAL TRIAL: NCT00423098
Title: A Randomized, Multicenter, Open-label, 6-month Study to Explore the Efficacy and Safety of Enteric-coated Mycophenolate Sodium in Combination With Two Corticosteroid Regimens for the Treatment of Lupus Nephritis Flare
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium in Combination With Two Corticosteroid Regimens for the Treatment of Lupus Nephritis Flare
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2420
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-05

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; enteric-coated mycophenolate sodium; EC-MPS; Myfortic
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Prednisone; Methylprednisolone

ARMS (2):
- Standard dose (Experimental): Mycophenolate sodium was administered orally in combination with a standard dose of corticosteroids (CS) administered as prednisone or prednisone equivalent (PRED). Mycophenolate sodium was administered in divided doses at a daily dose of 1440 mg during the first 2 weeks of the study and then at 2160 mg daily for the next 22 weeks. The dose of Prednisone was started at 1 mg per kg body weight and subsequently tapered according to the patient's weight. The planned treatment duration was 24 weeks.
  Interventions: Drug: Mycophenolate sodium; Drug: Prednisone; Drug: Methylprednisolone
- Low dose (Active Comparator): Mycophenolate sodium was administered in combination with a reduced dose of corticosteroids (CS) administered as prednisone or prednisone equivalent (PRED). Mycophenolate sodium was administered in divided doses at a daily dose of 1440 mg during the first 2 weeks of the study and then at 2160 mg daily for the next 22 weeks. The dose of Prednisone was started at 0.5 mg per kg body weight and subsequently tapered according to the patient's weight. The planned treatment duration was 24 weeks.
  Interventions: Drug: Mycophenolate sodium; Drug: Prednisone; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Mycophenolate sodium — Mycophenolate sodium as administered orally for 2 weeks at 1440mg daily and then increased to 2160mg daily for 22 weeks.
  Other Names: Myfortic
Drug: Prednisone — Oral prednisone or prednisone equivalent was started on Day 4 and subsequently tapered every 2 weeks according to the patient's weight.
Drug: Methylprednisolone — All patients received bolus therapy with 0.5 g of intravenous Methylprednisolone per day for 3 consecutive days.

SUMMARY:
The study will investigate the efficacy and safety of enteric-coated mycophenolate sodium in combination with two different corticosteroid (CS) regimes for the induction of remission of a lupus nephritis flare. Patients will be randomly allocated to standard CS regimen (group I) or to a reduced dose CS regimen (group II)

ELIGIBILITY:
Inclusion criteria

* Male or female patients with systemic lupus erythematosus (SLE)(at least 4 classification criteria)
* Aged ≥18 years,
* Proliferative lupus nephritis classified as ISN/RPS class III or IV
* Renal biopsy within the last 24-month preceding the study entry
* Proteinuria defined as >0.5 gram urine protein per gram urine creatinine at screening and baseline
* Clinical activity defined by one or more of the following changes in renal function: Serum creatinine >1.0 mg/dl (88.4 μmol/l)
* Microscopic hematuria defined as >5 red cells per high power field
* Presence of cellular casts

Exclusion criteria

* Patients with calculated creatinine clearance <30 ml/min (using the Cockcroft-Gault formula)
* Patients having received an intravenous (i.v.) corticosteroid bolus during the last 3 months,
* Patients having received oral or i.v. cyclophosphamide during the last 3 month
* Patients having received mycophenolate mofetil (MMF) within the preceding 3 months
* Use of any antibody therapy within the past 6 months
* Pregnant or nursing (lactating) women or women of child-bearing potential who are planning to become pregnant, or are not willing to use effective means of contraception throughout the study and during one month after the end of the study.
* Use of other investigational drugs within 1 month of enrollment (except for antibodies: within 6 months of enrollment
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures,
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Novartis, Bogotá, Colombia
- France (3):
  - Novartis, Créteil
  - Novartis, Nantes
  - Novartis Investigative Site, Paris
- Germany (2):
  - Novartis, Berlin
  - Novartis, Tübingen
- Novartis, Athens, Greece
- Hungary (2):
  - Novartis, Budapest
  - Novartis, Debrecen
- Italy (4):
  - Novartis, Brescia
  - Novartis, Ferrara
  - Novartis, Milan
  - Novartis, Padua
- Spain (2):
  - Novartis, Barcelona
  - Novartis, Madrid
- Novartis, Taichung, Taiwan
- Novartis, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose: Mycophenolate sodium was administered orally in combination with a standard dose of corticosteroids (CS) administered as prednisone or prednisone equivalent (PRED). Mycophenolate sodium was administered in divided doses at a daily dose of 1440 mg during the first 2 weeks of the study and then at 2160 mg daily for the next 22 weeks. The dose of CS was started at 1 mg per kg body weight and subsequently tapered according to the patient's weight. The planned treatment duration was 24 weeks.
- Low Dose: Mycophenolate sodium was administered orally in combination with a reduced dose of corticosteroids (CS) administered as prednisone or prednisone equivalent (PRED). Mycophenolate sodium was administered in divided doses at a daily dose of 1440 mg during the first 2 weeks of the study and then at 2160 mg daily for the next 22 weeks. The dose of CS was started at 0.5 mg per kg body weight and subsequently tapered according to the patient's weight. The planned treatment duration was 24 weeks.
Period: Overall Study
Arm/Group | Standard Dose | Low Dose
Started | 42 (Total number of patients screened was 90, but the total number of randomized patients was 81.) | 39
Completed | 39 (Completed 24 weeks of study medication.) | 35
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose | Low Dose | Total
Number analyzed (Participants) | 42 | 39 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.53) | 34.2 (10.74) | 33.1 (9.65)
Age, Customized [Number; unit: participants]
  18-29 years | 20 | 18 | 38
  30-39 years | 16 | 10 | 26
  40-49 years | 4 | 6 | 10
  50-59 years | 2 | 4 | 6
  >=60 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Remission
Description: Complete remission was defined as urine protein/urine creatinine ratio < 0.5 gram urine protein per gram urine creatinine, urine sediment normalized (no cellular casts, < 5 red cells per high power field), and serum creatinine within 10% of normal range according to local lab.
Time Frame: 24 Weeks
Population: Intention to treat (ITT) population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
Participants
  Yes | 8 | 8
  No | 34 | 31

2. Secondary Outcome: Number of Patients With Complete Remission
Description: Complete remission was defined as urine protein/urine creatinine ratio < 0.5 gram urine protein per gram urine creatinine, urine sediment normalized (no cellular casts, < 5 red cells per high power field), and serum creatinine within 10% of normal value.
Time Frame: 12 Weeks
Population: Intention to treat (ITT) population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
participants
  Yes | 9 | 5
  No | 33 | 34

3. Secondary Outcome: Number of Patients With Partial Remission
Description: Partial remission was defined as urine protein/creatinine ratio reduced by at least 50% from baseline and stable serum creatinine within 10% of baseline value) or improved.
Time Frame: Baseline to 12 and 24 weeks
Population: Intention to treat (ITT) population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
Participants
  At 12 weeks - Yes | 16 | 11
  At 12 weeks - No | 26 | 28
  At 24 weeks - Yes | 20 | 14
  At 24 weeks - No | 22 | 25

4. Secondary Outcome: Cumulative Dose of Prednisone Equivalent Corticosteroids (CS)
Description: Corticosteroid use was measured as cumulative dose until 12 and 24 weeks of treatment as well as daily doses at baseline, 12 and 24 weeks.
Time Frame: 12 Weeks and 24 Weeks
Population: Intention to treat (ITT) population: All randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
mg/kg
  Week 12 | 106.1 (13.55) | 68.2 (16.41)
  Week 24 | 114.2 (15.01) | 73.0 (17.76)

5. Secondary Outcome: Number of Patients With Moderate to Severe Flares
Description: A moderate to severe flare was defined as the occurrence of increased lupus activity after partial or complete remission, based on the presence of 1 BILAG A score or >=3 BILAG B scores. British Isles Lupus Assessment Group (BILAG) index divides lupus activity in 8 organs/systems which are each given a score of A to E. A=disease sufficiently active to need disease modifying treatment; B=problems requiring symptomatic treatment; C=mild stable disease; D=previously affected but currently inactive system; E=the system or organ has never been involved. BILAG score: A=9, B=3, C=1, D/E=0; range(0-72)
Time Frame: 12 and 24 weeks
Population: Intention to treat (ITT) population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
participants
  At week 12 - Yes | 0 | 0
  At week 12 - No | 42 | 39
  At week 24 - Yes | 1 | 0
  At week 24 - No | 41 | 39

6. Secondary Outcome: Duration of Exposure to Study Medication
Description: The duration of exposure was calculated as the date of the last Mycophenolate sodium dose minus the date of the last Mycophenolate sodium dose +1.
Time Frame: 24 weeks
Population: Safety population: All patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
days | 164.5 (24.87) | 157.7 (41.15)

7. Secondary Outcome: Number of Patients With Adverse Events and Infections
Description: Safety assessments included collecting all adverse events (AEs), serious adverse events (SAEs), with their severity and relationship to study drug. According to FDA 21CFR 314.80, a serious adverse event (SAE) is described as any adverse event that leads to death, is life threatening ( NIH criteria Grade 4), causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above.
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
participants
  At least one adverse event | 35 (5.63) | 30 (6.62)
  Any severe adverse event | 7 (7.08) | 3 (8.31)
  Any drug related adverse event | 18 (7.32) | 16 (8.35)
  Any serious adverse event | 8 | 4
  Any infection | 25 | 17
  Any severe infection | 3 | 1
  Any drug related infection | 10 | 6
  Any serious infection | 4 | 1

8. Secondary Outcome: Number of Patients With Treatment Failure
Description: Treatment failure was defined as no therapeutic response (without complete or partial remission) or premature discontinuation during the first 24 weeks from study medication or the study for any reason except complete or partial remission.
Time Frame: 12 Weeks and 24 Weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
participants
  At 12 weeks - Yes | 23 | 25
  At 12 weeks - No | 19 | 14
  At 24 weeks - Yes | 21 | 22
  At 24 weeks - No | 21 | 17

9. Secondary Outcome: Change From Baseline in Overall Disease Activity With Systematic Lupus Erythematosus Disease Activity Index (SLEDAI)
Description: SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index and was a well established global score index based on assessment of 24 items measuring a disease activity in the 10-day period prior to the assessment. SLEDAI item weights range from 1 for fever to 8 for seizures. A maximum theoretical score is 105. Total score range from 1 to 105. A flare has been defined as a SLEDAI score increase of 3 or more to a level of 8 or higher. During flares SLEDAI scores of 25 to 30 are common.
Time Frame: From Baseline to week 4, week 12 and week 24
Population: Intent-to-treat (ITT) population included all randomized patients who received at least one dose of study drug. Only patients with assessments at both baseline and post-baseline visits are summarized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
Units on a scale
  Change from Baseline to Week 4: (N= 39, 37) | -7.4 (5.63) | -7.7 (6.62)
  Change from Baseline to Week 12: (N= 41, 35) | -9.7 (7.08) | -10.3 (8.31)
  Change from Baseline to Week 24: (N= 39, 34) | -10.3 (7.32) | -9.8 (8.35)

10. Secondary Outcome: Change From Baseline in Overall Disease Activity With British Isles Lupus Assessment Group (BILAG)
Description: BILAG (British Isles Lupus Assessment Group) index divides lupus activity into 8 organs/systems and was based on the principle of the physician's intention to treat, assessing activity in the previous one month. Each organ or system was given a score of A to E, where A = disease that is sufficiently active to require disease modifying treatment; a B = problems requiring symptomatic treatment; C = stable mild disease; D = previously affected but currently inactive system; and E = the system or organ has never been involved. [A=9, B=3, C=1, D/E=0 the score range for each patient will be 0-72].
Time Frame: From Baseline to week 4, week 12 and week 24
Population: Intent-to-treat (ITT) populationincluded all randomized patients who received at least one dose of study drug. Only patients with assessments at both baseline and post-baseline visits are summarized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Standard Dose | Low Dose
Number analyzed (Participants) | 42 | 39
Units on a scale
  Change from baseline Week 4: (N= 40, 37) | -4.8 (5.34) | -5.5 (6.50)
  Change from baseline Week 12: (N= 41, 35) | -8.6 (6.76) | -8.7 (6.19)
  Change from baseline Week 24: (N= 40, 34) | -8.6 (5.79) | -9.4 (5.52)

ADVERSE EVENTS:
Arm/Group | Standard Dose | Low Dose
Serious Adverse Events (participants affected / at risk) | 8/42 | 4/39
Other Adverse Events (participants affected / at risk) | 28/42 | 18/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose (N=42) | Low Dose (N=39)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Epstein-barr virus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose (N=42) | Low Dose (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Gastritis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
Oedema peripheral (General disorders) | 4 | 5
Folliculitis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 6 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypertension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.